CLINICAL TRIAL: NCT05773911
Title: Treatment of Advanced Periodontitis Using an Oscillating Chitosan Device With or Without a Chitosan Gel - a Randomized Parallel Arm Clinical Trial
Brief Title: Treatment of Advanced Periodontitis With a Chitosan Brush and a Chitosan Gel
Acronym: Chitosangel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Caspar Wohlfahrt (Industry)
Collaborators: Dr Caspar Wohlfahrt (Unknown); Dr Maria Balta (Unknown)
Responsible Party: Sponsor-Investigator, Caspar Wohlfahrt, Head of Research and Development, Labrida AS
Organization: Labrida AS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 219125
Record Dates: First submitted 2022-09-15; First posted 2023-03-17 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Periodontitis; Periodontal Pocket; Periodontal Diseases; Periodontal Inflammation
Keywords: Periodontitis; Periodontal disease; Periodontal pocket
MeSH Terms: conditions — Periodontitis; Periodontal Pocket; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: This efficacy study will be a prospective multicenter parallel arm, examiner blinded, randomized clinical trial of 12 months' duration.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Curettes+ Ultrasonic scalers supragingivally and a chitosan brush in oscillating handpiece subgingivally with adjunct 4% chitosan gel (pH 3.48).
  Interventions: Device: 4% chitosan gel (pH 3.48).
- Control (Active Comparator): Curettes+ Ultrasonic scalers supragingivally and a chitosan brush in oscillating handpiece subgingivally
  Interventions: Device: Reciprocal Chitosan brush

INTERVENTIONS:
Device: 4% chitosan gel (pH 3.48). — Reciprocal Chitosan brush with 4% chitosan gel (pH 3.48).
  Other Names: Gelix
  Arms: Test
Device: Reciprocal Chitosan brush — Reciprocal Chitosan brush
  Other Names: Labrida BioClean
  Arms: Control

SUMMARY:
In the here suggested study, the aim is to test non-surgical treatment of advanced periodontal disease with a chitosan brush with or without chitosan gel in patients with advanced periodontal disease having responded poorly to a more conventional treatment strategy, with the aim to hinder the progression of bone loss around the teeth.

DETAILED DESCRIPTION:
Labrida GeliX Chitosan gel 4% (LABRIDA AS, Oslo, Norway) is a chitosan gel. Labrida GeliX Chitosan gel 4% consists of water, chitosan (4%) and lactic acid (2%) and with pH 3.86. In this study GeliX Chitosan gel 4% shall be tested as an adjunct to mechanical debridement of infected tooth surfaces affected by periodontal disease and which have responded poorly to conventional treatment.

Hypotheses and study objectives

Null hypothesis and alternate hypothesis

H0:

There will be no significant difference in reduction in parameters of periodontal inflammation between the test and control groups after 6 and 12 months.

HA:

There will be a significant difference in reduction in parameters of periodontal inflammation between the test and control groups after 6 and 12 months.

Primary Objective Difference between test and control groups in change in inflammation tested by measuring the surrogate markers Pocket Probing Depth (PPD) and Bleeding on Probing (BoP) This will be done to assess the clinical efficacy of Labrida GeliX Chitosan gel 4% used in combination with Labrida BioClean® for treatment of advanced periodontal disease (2017 World Workshop Stage III and IV Grade B) Primary endpoint is reduction in periodontal disease as measured clinically up to three months after therapy.

Secondary Objectives • Difference between test and control groups in change in periodontal attachment loss tested by measuring clinical attachment loss (CAL) and bone level differences on radiographs at baseline and 6 and 12 months. This will be done to assess safety of Labrida GeliX Chitosan gel 4% used in combination with Labrida BioClean®, by evaluating the occurrence of adverse events.

Design of clinical investigation

This efficacy study will be a prospective multicenter parallel arm, examiner blinded, randomized clinical trial of 12 months' duration.

Patient screening, inclusions and all clinical examinations will be performed by a board-certified specialist in periodontology at the test centers. Treatment will be performed by a registered separate therapist, either dentist or dental hygienist.

Clinical variables of periodontal disease will be recorded at baseline, 1 week, 4 weeks and at 3, 6, 9 and 12 months. Radiographs will be taken at baseline and at 6 and 12 months. Treatment will be performed at baseline and thereafter at three months intervals.

Follow-up

* Intraoral radiographs will be taken at baseline and at 6 months to exclude progression in bone loss.
* Post clinical data 4 weeks after treatment and 3, 6, and 9 months after treatment.

Objectives

Primary:

Primary endpoint is reduction in periodontal disease as measured clinically up to three months after therapy.

Secondary:

• Evaluation of difference between test and control groups in change in periodontal attachment loss tested by measuring clinical attachment loss (CAL) and bone level differences on radiographs at baseline and 6 and 12 months.

Study financing The study is financed by the sponsor Labrida AS.

Enrollment and Randomization

Patients will be allocated to one of the following two treatments:

A) C+ USS supragingivally and a chitosan brush in oscillating handpiece subgingivally and irrigation with sterile saline B) C+ USS supragingivally and a chitosan brush in oscillating handpiece subgingivally with adjunct 4% chitosan gel (pH 3.86) and irrigation with sterile saline followed by application of chitosan gel in the pockets.

A computer-generated block randomization will be used to ensure equal sample sizes.

Labrida GeliX Chitosan gel 4% used as an adjunct to non-surgical treatment with Labrida BioClean® is the investigational device while the comparator in the control group is Labrida BioClean® alone (CE 2460). No other device or medication will be used in the trial.

Subjects Target population In the here suggested study, the aim is to test non-surgical treatment of advanced periodontal disease with a chitosan brush with or without chitosan gel in patients with advanced periodontal disease having responded poorly to a more conventional treatment strategy, with the aim to hinder the progression of bone loss around the teeth.

Main inclusion criteria Patients with at least 3 teeth but less than 8 teeth with advanced periodontal attachment loss (2017 World Workshop Stage III and IV Grade B), Clinical Attachment Loss (CAL) ≥5 mm, probing pocket depth (PPD) ≥5mm and ≤8 mm and inflammation as demonstrated by a modified Bleeding on Probing (BoP) grade 2 (line) or 3 ("spontaneous").

Total expected duration of the clinical investigation Study period Q2 2023 until Q2 2024 Expected duration of each subject participation 12 months

Patients 40 patients diagnosed with advanced periodontitis will be included. 20 patients will be treated with the control treatment (the chitosan brush), 20 patients will be treated with the test treatment (chitosan brush with chitosan gel).

Details of measures to be taken to minimize bias Bias will be avoided through double blinding and randomization. Confounding factors will be avoided through inclusion criteria and randomization.

Clinical procedures and diagnostic methods

Preoperative evaluation Clinical and radiographic evaluation including periodontal and general dental status. The radiographic evaluation includes intraoral radiography with apical radiographs and vertical bitewings on molars and premolars. Clinical screening includes routine history and physical examination, admission criteria, signed informed consent and pain assessments.

The full-mouth plaque index using dichotomous scoring shall be below 20% prior to final inclusion.

Clinical procedure 1) Full mouth supragingival debridement to remove supragingival visual calculus will be performed with hand curettes and ultrasonic scaler

Subgingival debridement after randomization to test or control group:

2 A) Control group: The periodontal pockets in the patients in the control group will be treated with C+ USS supragingivally and a chitosan brush in an oscillating handpiece (NSK ER10 + TEQ-Y) subgingivally for 2 minutes. Thereafter irrigation using sterile saline.

2 B) Test group: The periodontal pockets in the patients in the test group will be treated with C+ USS supragingivally and a chitosan brush in oscillating handpiece subgingivally with adjunct 4% chitosan gel subgingivally (pH 3.86) and irrigation using sterile saline. and application of the chitosan gel into the pockets A computer-generated block randomization will be used to ensure equal sample sizes.

The treatments will be repeated every three months and the terminal examination will be at 12 months. All treatments will be performed by a registered dental hygienist. All examinations will be performed by a board certified periodontist other than the sponsor. The sponsor representative will not have an active role in the study other than screening of patients and monitoring of the study.

Prophylaxis Endodontic lesions, prosthetic complications and dental decay should be treated before study start. Plaque Index (dichotomous scoring) should be ≤20%.

Examinations Medical history will be carefully recorded prior to examination. Clinical variables of inflammation will be measured at baseline and 4 weeks, 12 weeks 6, 9 and 12 months after baseline.

Non-invasive sampling of gingival crevicular fluid from the tooth crevice at baseline and one and 4 weeks will be undertaken and used for analysis of changes in inflammatory markers after treatment.

Probing pocket depths will be recorded at 6 sites (mesio-buccally, buccaly, disto-buccally, disto-palataly, palataly, mesio-palataly) around each included tooth using a regular periodontal probe according to the examiner's preferences. Bleeding on probing at the included sites will be assessed using a three-graded index within 30 seconds following probing of the pocket using a modified bleeding on probing index (mBoP) (28). Suppuration at the included sites will be recorded using dichotomous scoring. CAL (ECJ to base of pocket) will be recorded at 6 sites per included tooth at baseline and at 6 and 12 months. Furcations will be recorded (Hampf 0, I, II, III). Mobility will be recorded (Miller 0,1,2,3). Plaque at the included teeth and for the full dentition, will also be assessed using dichotomous scoring. Radiographs will be taken at baseline and at 12 months.

Copies of informed consents and radiographs will be stored at each center, according to GCP - guidelines.

Routine history and physical examination will be performed, and information recorded in the Preoperative Patient History Record. The therapist may use his/her customary history and physical procedures; however, all data specified on the Preoperative Patient History Record will be recorded in the Case Report Form (CRF). Exclusion Criteria are also included in the form. Entries checked YES will exclude patients from admission into the study.

Peroperative procedures (At the time of the treatment) Treatment approach and technique will be carried out according to a standardized procedure agreed upon between the participating therapists.

POSTOPERATIVE FOLLOW-UP PROCEDURES All postoperative evaluations (Clinical examination (CAL, PLI, BoP, PPD, pus)) will be recorded on regular patient record and later transferred to the Case Report Form. Furthermore, intraoral radiographs will be taken at baseline and at 6 months to exclude progression in bone loss.

Clinical complications such as infection, pain etc. will be recorded during all postoperative follow-up visits, should they occur.

The GCF samples will be stored in a dedicated project biobank at the Institute of oral biology (Dr Maria Balta will be responsible for the project biobank) until all patients has undergone the 4 weeks control and thereafter sent to University of Minnesota, USA for Mass spectrometry-based metabolomics analysis of changes in some metabolites involved in the inflammation and treatment response between baseline and 1 week and 4 weeks. A wide range of metabolites involved in the inflammatory response will be included in the analyses. Metabolites involved in degradation of chitosan will also be analysed for. Professor Massimo Costalonga, University of Minnesota will be responsible for the analyses. Any remaining biologic material will be destroyed.

Statistical consideration Sample size If a PPD difference in the change of PPD between methods of 1 mm is to be detected at a=0.05 and a power of = 0.2, the appropriate number of subjects per group would be 20. Hence, the inclusion of 40 subjects in the study would yield the necessary statistical power.

Statistical evaluation After completion of the study, the statistical analysis will be performed by the principal investigators in collaboration with a biostatistician.

A two-sided statistical test will be used since both positive and potential negative outcomes will be evaluated. Sigma Stat will be used. All data will be transferred from the CRF to Sigma Stat files. The statistical computations will be cross checked with a professional biostatistician.

The report will form the basis for the Clinical Investigation Report and a manuscript intended for publication in a dental peer reviewed scientific journal.

Ethics Committee Approval The study has been accepted by the Regional Ethical Review board

.

ELIGIBILITY:
Inclusion criteria:

Patients with at least 3 teeth but less than 8 teeth with advanced periodontal attachment loss.

Clinical Attachment Loss (CAL) ≥5 mm, probing pocket depth (PPD) ≥5mm and ≤8 mm and inflammation as demonstrated by a modified Bleeding on Probing (BoP) grade 2 (line) or 3 ("spontaneous").

Exclusion criteria:

* Ongoing radiotherapy, ongoing chemotherapy, pregnant or nursing patients, prosthetic factors making access to clinical measurements impossible
* Poor oral hygiene with plaque at >20% of the surfaces
* Periodontal pockets reaching to the apex of teeth.
* Teeth with active peri-apical pathology
* Teeth with root resorption as seen on radiographs
* Teeth with prosthodontic technical complications should be excluded or treated before inclusion (e.g., overhangs, open contacts with food impaction)
* Teeth with pockets from other reasons than periodontal disease
* Teeth with traumatic occlusion should be excluded or treated before inclusion (i.e., fremitus)
* Patients diagnosed with Periodontal disease grade C i.e., rapid rate of progression
* Sites in direct proximity with site(s) where patient places snuff (Copenhagen) will be excluded

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pocket Probing depths change | 12 months
  Difference between test and control sites in Probing Pocket Depth (PPD)4 weeks , 3 months, 6, 9 and 12 months after baseline.
Bleeding on Probing change | 12 months
  Change in periodontal inflammation measured with the inflammation surrogate marker Bleeding on Probing using a categorial scale (modified Bleeding on Probing index (mBoP: 0, 1, 2, 3)) and

CONTACTS AND LOCATIONS:
Locations (1):
- Bjerke tannmedisin, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein O, Balta MG, Wohlfahrt JC. Treatment of Residual Pockets in Stage III and IV Periodontitis Using an Oscillating Chitosan Device With or Without a Chitosan Gel-A Randomised Parallel-Arms Clinical Trial. J Clin Periodontol. 2026 Jan 22. doi: 10.1111/jcpe.70086. Online ahead of print. PMID 41568740